CLINICAL TRIAL: NCT00123058
Title: Take Control of Your Blood Pressure (TCYB)
Brief Title: Comparison of Two Programs to Improve Blood Pressure Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00005845; R01HL070713 (NIH); NCT00129103 (obsolete NCT alias)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
Keywords: Hypertension; Cariovascular Diseases; Health Illiteracy
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension | interventions — Blood Pressure Monitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Nurse administered (Experimental): Nurse Administered Intervention:
  Subject received nurse administered behavioral intervention every 8 weeks via telephone for 24 months.
  Interventions: Behavioral: Nurse administered
- Nurse & BP monitor (Experimental): Subjects received both a nurse administered behavioral intervention via telephone every 8 weeks for 24 months and a study provided home BP monitor. Subject recorded home BP 3 times per week for 24 months.
  Interventions: Behavioral: Nurse administered; Device: BP Monitor
- Usual Care (No Intervention): Subjects received neither home BP monitor nor nurse phone intervention.
- Home BP Monitor (Experimental): Subject received study provided home BP monitor. Subject recorded home BP 3 times per week for 24 months.
  Interventions: Device: BP Monitor

INTERVENTIONS:
Behavioral: Nurse administered — Subjects received a nurse administered behavioral intervention via telephone every 8 weeks for 24 months.
  Arms: Nurse & BP monitor; Nurse administered
Device: BP Monitor — Subjects received a study provided home BP monitor and recorded home BP 3 times per week for 24 months.
  Arms: Home BP Monitor; Nurse & BP monitor

SUMMARY:
The purpose of this study is to improve adherence to blood pressure (BP) monitoring and medication compliance in individuals with high BP.

DETAILED DESCRIPTION:
BACKGROUND:

High BP is a major health problem, which contributes to high levels of morbidity and mortality. Elevated BP levels are a major risk factor for stroke, coronary artery disease (CAD), congestive heart failure (CHF), and kidney disease. In the United States, stroke rates are no longer improving and CHF and kidney failure rates continue to increase. Despite the availability of effective treatment, only 25% of individuals with high BP are able to control it effectively. The reasons for poor BP control vary; however, a predominant reason is poor adherence to medication instructions and life-style modification recommendations. This study will address these two sources of poor BP control through a real world, multifaceted approach.

DESIGN NARRATIVE:

This study will compare a nurse-administered tailored program to a home BP monitoring program to evaluate the impact each program has on BP control. The 5-year randomized controlled study will take place in a primary care setting and will enroll individuals with high BP. The nurse-administered program will be based on the principles of the Health Decision Model and will be designed to increase awareness, yet be easily integrated into the participant's medical care so as to enhance adherence with the prescribed treatment. The use of home BP monitors has been found to be associated with increased self management, medication adherence, and improved BP control.

Five hundred seventy individuals with high BP from two primary care clinics will be randomly assigned to receive either the nurse-administered program, home BP monitoring program, both programs, or regular medical care. Based on an initial assessment, participants assigned to the nurse-administered program will be involved in a behavioral education telephone program to promote medication adherence. This program will include support, reminders, and information on the risks of high BP, health behaviors, patient/doctor communication, literacy, and side effects. Participants will receive continuous education and will be monitored and supported to enhance medication adherence. Participants assigned to the home BP monitors will record their BP every other day and mail the results to the study physicians. The primary outcome will be whether or not the participant's BP is greater than 140/90 mm Hg (for non-diabetic individuals) or greater than 130/85 mm Hg (for diabetic individuals) at 6-month intervals over 24 months (5 total measurements). Descriptive statistics will be computed for all study variables stratified by treatment group. Because each participant may have a different number of measurements, the study physicians will model the responses and evaluate the programs using a mixed effects model for dichotomous outcomes. Based upon preliminary data, this study will improve participants' management of high BP, decrease health care utilization, and subsequently improve BP control.

Additionally, a subset (n=250) of those enrolled and randomized to either the nurse administered program or usual care will be evaluated separately on the programs's effect on both primary (blood pressure control) and secondary outcome measures (changes in hypertension risk perception,satisfaction with care, patient confidence following recommended regimen, and self-reported adherence to recommended regimens.) Masking for this is open label.

ELIGIBILITY:
Inclusion Criteria:

* Visited Duke General Internal Medicine Primary Care Clinic at Pickett Road or Duke Outpatient Clinic between April 2003 and April 2004
* Diagnosed with high BP
* Currently residing in an eight county area, including Durham County, NC and surrounding counties
* Currently taking BP medication
* Receives most medical care at the Duke Primary Care clinics
* Able to speak and understand English over the phone

Exclusion Criteria:

* Diagnosed with dementia
* Diagnosed with Parkinson's Disease
* Diagnosed with atrial fibrillation
* Diagnosed with end stage kidney disease
* Hospitalized for stroke, heart attack, or coronary artery revascularization in the 3 months prior to study entry
* Diagnosed with metastatic cancer in the 3 months prior to study entry
* Receiving kidney dialysis
* Pregnant or expecting to become pregnant in the 2 years following study entry
* Currently residing in a nursing home or receiving home health care
* Severely impaired speech or hearing
* Participating in another blood pressure study
* Has another family member participating in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2003-06; Primary Completion 2005-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
BP measurement | Measured at 6 months

SECONDARY OUTCOMES:
Satisfaction with care | Measured at 6 and 24 months
Risk associated with hypertension | Measured at 6 and 24 months
Self reported adherence | Measured at 6 and 24 months
Efficacy with treatment | Measured at 6 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B. Bosworth, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Bosworth HB, Olsen MK, Gentry P, Orr M, Dudley T, McCant F, Oddone EZ. Nurse administered telephone intervention for blood pressure control: a patient-tailored multifactorial intervention. Patient Educ Couns. 2005 Apr;57(1):5-14. doi: 10.1016/j.pec.2004.03.011. PMID 15797147
- [Background] Hong TB, Oddone EZ, Dudley TK, Bosworth HB. Subjective and objective evaluations of health among middle-aged and older veterans with hypertension. J Aging Health. 2005 Oct;17(5):592-608. doi: 10.1177/0898264305279780. PMID 16177452
- [Background] Kim JW, Bosworth HB, Voils CI, Olsen M, Dudley T, Gribbin M, Adams M, Oddone EZ. How well do clinic-based blood pressure measurements agree with the mercury standard? J Gen Intern Med. 2005 Jul;20(7):647-9. doi: 10.1111/j.1525-1497.2005.0105.x. PMID 16050862
- [Background] Hong TB, Franks MM, Gonzalez R, Keteyian SJ, Franklin BA, Artinian NT. A dyadic investigation of exercise support between cardiac patients and their spouses. Health Psychol. 2005 Jul;24(4):430-4. doi: 10.1037/0278-6133.24.4.430. PMID 16045379
- [Background] Bosworth HB, Olsen MK, Oddone EZ. Improving blood pressure control by tailored feedback to patients and clinicians. Am Heart J. 2005 May;149(5):795-803. doi: 10.1016/j.ahj.2005.01.039. No abstract available. PMID 15894959
- [Background] Bosworth HB, Bartash RM, Olsen MK, Steffens DC. The association of psychosocial factors and depression with hypertension among older adults. Int J Geriatr Psychiatry. 2003 Dec;18(12):1142-8. doi: 10.1002/gps.1026. PMID 14677147
- [Background] Trivedi RB, Ayotte B, Edelman D, Bosworth HB. The association of emotional well-being and marital status with treatment adherence among patients with hypertension. J Behav Med. 2008 Dec;31(6):489-97. doi: 10.1007/s10865-008-9173-4. Epub 2008 Sep 9. PMID 18780175
- [Background] Bosworth HB, Powers B, Grubber JM, Thorpe CT, Olsen MK, Orr M, Oddone EZ. Racial differences in blood pressure control: potential explanatory factors. J Gen Intern Med. 2008 May;23(5):692-8. doi: 10.1007/s11606-008-0547-7. Epub 2008 Feb 21. PMID 18288540
- [Background] Powers BJ, Oddone EZ, Grubber JM, Olsen MK, Bosworth HB. Perceived and actual stroke risk among men with hypertension. J Clin Hypertens (Greenwich). 2008 Apr;10(4):287-94. doi: 10.1111/j.1751-7176.2008.07797.x. PMID 18401226
- [Background] Ayotte BJ, Allaire JC, Bosworth H. The associations of patient demographic characteristics and health information recall: the mediating role of health literacy. Neuropsychol Dev Cogn B Aging Neuropsychol Cogn. 2009 Jul;16(4):419-32. doi: 10.1080/13825580902741336. Epub 2009 May 8. PMID 19424920
- [Background] Voils CI, Sandelowski M, Dahm P, Blouin R, Bosworth HB, Oddone EZ, Steinhauser KE. Selective adherence to antihypertensive medications as a patient-driven means to preserving sexual potency. Patient Prefer Adherence. 2008 Feb 2;2:201-6. doi: 10.2147/ppa.s3796. PMID 19920964
- [Background] Reed SD, Li Y, Oddone EZ, Neary AM, Orr MM, Grubber JM, Graham FL, Olsen MK, Svetkey LP, Dolor RJ, Powers BJ, Adams MB, Bosworth HB. Economic evaluation of home blood pressure monitoring with or without telephonic behavioral self-management in patients with hypertension. Am J Hypertens. 2010 Feb;23(2):142-8. doi: 10.1038/ajh.2009.215. Epub 2009 Nov 19. PMID 19927132
- [Background] Trivedi RB, Ayotte BJ, Thorpe CT, Edelman D, Bosworth HB. Is there a nonadherent subtype of hypertensive patient? A latent class analysis approach. Patient Prefer Adherence. 2010 Jul 21;4:255-62. doi: 10.2147/ppa.s11335. PMID 20694185
- [Result] Bosworth HB, Olsen MK, Dudley T, Orr M, Neary A, Harrelson M, Adams M, Svetkey LP, Dolor RJ, Oddone EZ. The Take Control of Your Blood pressure (TCYB) study: study design and methodology. Contemp Clin Trials. 2007 Jan;28(1):33-47. doi: 10.1016/j.cct.2006.08.006. Epub 2006 Aug 16. PMID 16996808
- [Result] Bosworth HB, Olsen MK, Neary A, Orr M, Grubber J, Svetkey L, Adams M, Oddone EZ. Take Control of Your Blood Pressure (TCYB) study: a multifactorial tailored behavioral and educational intervention for achieving blood pressure control. Patient Educ Couns. 2008 Mar;70(3):338-47. doi: 10.1016/j.pec.2007.11.014. Epub 2007 Dec 31. PMID 18164894
- [Derived] Muir KW, Grubber J, Mruthyunjaya P, McCant F, Bosworth HB. Progression of diabetic retinopathy in the hypertension intervention nurse telemedicine study. JAMA Ophthalmol. 2013 Jul;131(7):957-8. doi: 10.1001/jamaophthalmol.2013.81. No abstract available. PMID 23702951
- [Derived] Bosworth HB, Olsen MK, Grubber JM, Neary AM, Orr MM, Powers BJ, Adams MB, Svetkey LP, Reed SD, Li Y, Dolor RJ, Oddone EZ. Two self-management interventions to improve hypertension control: a randomized trial. Ann Intern Med. 2009 Nov 17;151(10):687-95. doi: 10.7326/0003-4819-151-10-200911170-00148. PMID 19920269